CLINICAL TRIAL: NCT06164132
Title: The Pivotal Influence of Obesity on Body Composition and Ovarian Doppler in Different Polycystic Ovarian Syndrome Phenotypes: An Observational Study
Brief Title: Pivotal Influence of Obesity on Body Composition and Ovarian Doppler in Different Polycystic Ovarian Syndrome Phenotypes
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Helwan University (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant Professor, Cairo University
Other Study IDs: P.T.REC/012/004609
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome; Obesity
Keywords: Polycystic Ovary Syndrome; Obesity; Body composition; Ovarian Doppler
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Weight group: Their BMI ranged from 18.5 to 24.9 kg/m2.
  Interventions: Other: Evaluation
- Overweight group: Their BMI ranged from 25 to 29.9 kg/m2.
  Interventions: Other: Evaluation
- Obese group: Their BMI was ≥ 30 kg/m2.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Evaluation through PCOS Phenotypes, measurements of Body weight, height, waist and hip circumferences, Dual-energy X-ray absorptiometry, and Sonographic examination.

SUMMARY:
The study aimed to explore the impact of obesity on both body composition and ovarian Doppler parameters across various phenotypes of females diagnosed with polycystic ovarian syndrome (PCOS). Additionally, the investigation seeked to establish correlations between these parameters and their prevalence concerning the clinical criteria of PCOS.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is a complex and multifactorial condition characterized by endocrinological, reproductive, metabolic, and biochemical abnormalities, affecting 12% to 21% of reproductive-aged females. It has emerged as a significant global public health concern. However, variations in diagnostic criteria and patient selection have led to considerable discrepancies in the absolute prevalence of PCOS and its temporal trends. Previous studies have examined ovarian volume and blood flow indices in both obese and non-obese females with PCOS, albeit employing different criteria for obesity classification. Notably, none have compared these parameters across normal weight, overweight, and obese PCOS females. Therefore, the current study aims to explore the impact of obesity on body composition and ovarian Doppler parameters within distinct PCOS phenotypes. An additional objective is to assess correlations between anthropometric, body composition, and ovarian Doppler parameters and the prevalence of PCOS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 18 to 40 years old.
* Individuals with Polycystic Ovary Syndrome (PCOS) should exhibit at least two of the three features outlined in the Rotterdam criteria for diagnosis, encompassing oligo- or anovulation, clinical and/or biochemical indications of hyperandrogenism, and the presence of polycystic ovaries as identified through ultrasonography.

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Thyroid dysfunction
* Hyperprolactinemia
* Androgen-secreting tumors
* Cushing syndrome
* Undergoing any medical therapy for the treatment of PCOS or for weight loss.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: They were recruited from the gynecology and infertility clinic, for Doppler sonographic examination and body composition analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Phenotypes of PCOS | 4 months
  The patients were categorized into four distinct phenotypes: Type I, characterized by oligomenorrhea/amenorrhea and hyperandrogenism (O+H); Type II, exhibiting polycystic ovaries and hyperandrogenism (P+H); Type III, featuring oligomenorrhea/amenorrhea and polycystic ovaries (O+P); and Type IV, presenting with oligomenorrhea/amenorrhea, polycystic ovaries, and hyperandrogenism (O+P+H).
Body mass index (BMI) | 4 months
  The height and weight were determined for each female in the three groups to calculate her BMI = (weight in kg)/(height in m2)
Waist hip ratio (WHR) | 4 months
  The waist and hip circumferences were taken for each female in the three groups for calculating waist and hip ratio (WHR) by dividing waist circumference (WC) on the hip circumference (HC).
Total and regional fat mass | 4 months
  They were measured by Dual-energy X-ray absorptiometry.
Total and regional lean mass | 4 months
  They were measured by Dual-energy X-ray absorptiometry.
Ovarian volume | 4 months
  The ovarian volume was computed utilizing the ellipsoid formula, which involves multiplying the dimensions of length, width, and height by a constant factor of 0.523.
Peak systolic velocity (PSV) | 4 months
  It was recorded for each female in the three groups by Color Doppler ultrasound.
End diastolic velocity (EDV) | 4 months
  It was recorded for each female in the three groups by Color Doppler ultrasound.
Resistive index (RI) | 4 months
  The Resistance Index (RI) was determined by dividing the difference between Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) by PSV. A lower value of RI is indicative of increased blood flow
Pulsatility index (PI) | 4 months
  The Pulsatility Index (PI) was calculated by dividing the difference between Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) by the mean maximum flow velocity. A reduced PI value is indicative of heightened blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Safenaz Y. El Sherity, Assis. Prof., Principal Investigator — National Research Centre, Egypt
Locations (1):
- Cairo University, Giza, Egypt